CLINICAL TRIAL: NCT00631787
Title: Evaluation of Systemic Toxicity Associated With Allogeneic Peripheral Blood Stem Cell Infusion
Brief Title: Evaluation of Toxicity From Stem Cell Transplant
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 080084; 08-H-0084
Record Dates: First submitted 2008-03-07; First posted 2008-03-10 (Estimated); Last update posted 2019-06-17 (Actual); Status verified 2015-12-07

CONDITIONS: Organ Dysfunction; Hemolysis
Keywords: Nitric Oxide; Hemolysis; Plasma Hemoglobin; Dimethyl Sulfoxide; Organ Dysfuntion; Healthy Volunteer; HV
MeSH Terms: conditions — Hemolysis

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This study will try to determine what causes toxic side effects of stem cell transplantation, such as increased blood pressure, increased heart rate, decreased kidney function and abnormal heart rhythms. Stem cells are used to treat various diseases, including cancer, aplastic anemia and sickle cell disease. The cells may be given fresh to the patient or they may be preserved first with a chemical called DMSO and frozen for later use. Some stem cell transplant procedures include infusion of red blood cells along with the stem cells. This study will examine whether side effects of stem cell transplants are associated with the DMSO preservative in frozen cells or with hemoglobin (a protein released from defrosted red blood cells) or neither of these factors.

Healthy volunteers and patients scheduled to receive a stem cell transplant may be eligible for this study. Candidates must be between 10 and 80 years of age.

Transplant patients will undergo a stem cell transplant. The cells are infused through a catheter placed in a vein for the procedure. Depending on the patient s requirements, the infusion may or may not include red blood cells and may or may not contain DMSO. Healthy volunteers undergo a 4-hour saline infusion. The saline (water mixed with salt) is infused through a catheter (plastic tube) placed in a vein in the arm. In addition, all participants have the following tests and procedures:

* Heart monitoring: Healthy volunteers wear a portable heart monitor, attached to the chest using four stickers, for 24 hours starting the morning of the infusion. Transplant patients wear the same device for 48 hours, starting the morning before the infusion.
* Blood draws and urine collections before, during, just after and the morning after the infusion of saline or stem cells.
* Heart ultrasound before, during or just after and the morning after the infusion.
* Peripheral artery tonometry: A small cup is placed on one finger of each hand to measure blood flow in the finger. A blood pressure cuff is inflated around the lower arm and tight pressure is maintained for about 5 minutes.

DETAILED DESCRIPTION:
Allogeneic and autologous bone marrow transplantation is currently the only curative option for many patients with life-threatening hematologic illnesses and malignancies. Peripheral blood stem cell (PBSC) infusion has been associated with systemic toxicities including arrhythmias, hypertension, and organ dysfunction. It has been thought that the preservative dimethyl sulfoxide (DMSO) that is frequently used to store frozen PBSCs may be the etiology of the adverse effects that occur during the infusion. However, we hypothesize that the red blood cells that rupture upon thawing infused with the graft release free hemoglobin which scavenges nitric oxide. This can lead to systemic vasoconstriction and organ dysfunction. In this protocol, we will monitor subjects who are undergoing PBSC transplantation with either fresh grafts that lack DMSO or frozen whole grafts. We will also evaluate patients who receive purified stem cell grafts, which will contain negligible red blood cells and associated free hemoglobin. We will then measure the frequency of infusion-related systemic toxicity and organ dysfunction between the groups.

ELIGIBILITY:
* INCLUSION CRITERIA HEALTHY VOLUNTEERS:

Ages 10 to 80

Normal renal function: creatinine less than 1.5 mg/dL in subjects greater than or equal to 18 years of age, less than or equal to 1.0 mg/dL in subjects 13 to 17 years of age, less than or equal to 0.7 in subjects 10 to 12 years of age, and proteinuria less than 1+

Normal liver function: bilirubin less than 1.5 mg/dL and transaminases within normal limits

Normal pulmonary arterial pressure by transthoracic echocardiogram (tricuspid regurgitant velocity less than 2.5 m/s)

Ability to comprehend and willing to sign an informed consent/assent

INCLUSION CRITERIA ALL OTHERS:

Ages 10-80

Otherwise as stated on the subject s primary protocol

EXCLUSION CRITERIA HEALTHY VOLUNTEERS:

History of clinically significant cardiac or pulmonary disease

EXCLUSION CRITERIA ALL OTHERS:

Patients receiving nitrate antihypertensive medications

Clinically unstable patients in which transfer to the intensive care unit is being considered

Otherwise as stated on the subject s primary protocol

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2008-02-29; Study Completion 2015-12-07

CONTACTS AND LOCATIONS:
Overall Officials: Courtney D Fitzhugh, M.D., Principal Investigator — National Heart, Lung, and Blood Institute (NHLBI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Kessinger A, Schmit-Pokorny K, Smith D, Armitage J. Cryopreservation and infusion of autologous peripheral blood stem cells. Bone Marrow Transplant. 1990 Jan;5 Suppl 1:25-7. No abstract available. PMID 1969303
- [Background] Styler MJ, Topolsky DL, Crilley PA, Covalesky V, Bryan R, Bulova S, Brodsky I. Transient high grade heart block following autologous bone marrow infusion. Bone Marrow Transplant. 1992 Nov;10(5):435-8. PMID 1464006
- [Background] Keung YK, Lau S, Elkayam U, Chen SC, Douer D. Cardiac arrhythmia after infusion of cryopreserved stem cells. Bone Marrow Transplant. 1994 Sep;14(3):363-7. PMID 7994256
- [Derived] Fitzhugh CD, Unno H, Hathaway V, Coles WA, Link ME, Weitzel RP, Zhao X, Wright EC, Stroncek DF, Kato GJ, Hsieh MM, Tisdale JF. Infusion of hemolyzed red blood cells within peripheral blood stem cell grafts in patients with and without sickle cell disease. Blood. 2012 Jun 14;119(24):5671-3. doi: 10.1182/blood-2011-11-392654. Epub 2012 Apr 30. PMID 22547579